CLINICAL TRIAL: NCT00739115
Title: The Use of Heliox Via Nasal CPAP to Prevent Early CPAP Failure in Premature Infants: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawaii Pacific Health (Other)
Collaborators: Hawaii Community Foundation (Other); Hawaii Medical Service Association (Other)
Responsible Party: Principal Investigator, Charles R. Neal,, Professor, Hawaii Pacific Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-026-1-HPH1
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: Respiratory; Distress; Prematurity; Heliox; CPAP
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Heliox gas added to nasal CPAP for the first 72 hours of life
  Interventions: Other: Heliox gas
- 2 (No Intervention): Conventional nasal CPAP for the first 72 hours of life

INTERVENTIONS:
Other: Heliox gas — Heliox gas used in conjunction with nasal CPAP
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the safety and utility of using heliox gas in combination with nasal CPAP in premature infants. The investigators hypothesize that using heliox gas in combination with nasal CPAP will results in decreased early nasal CPAP failure requiring intubation and mechanical ventilation.

DETAILED DESCRIPTION:
Introduction: In recent years there has been an increased use of nasal continuous positive airway pressure (nCPAP) in the management of premature infants with respiratory distress syndrome (RDS). The use of early nCPAP eliminates the need for endotracheal intubation and mechanical ventilation, and their associated morbidities. In clinical practice a significant number of extremely low birth weight (ELBW) infants with RDS fail nCPAP therapy within the first 72 hours of life and require rescue endotracheal intubation. The clinical factors resulting in nCPAP failure are hypoxemia, hypoventilation, muscular fatigue and/or apnea. Helium is a biologically inert gas that is used in medicine as a carrier for oxygen. Heliox (mixture of helium and oxygen) has been used safely in neonates for decades and its use has been consistently been shown to improve oxygenation, enhance ventilation and decrease the work of breathing. Prior studies using heliox in the management of premature infants with RDS have shown clear therapeutic benefits. The use of heliox delivered via a nCPAP device (Hx-nCPAP) has recently been reported in infants with bronchiolitis. Given the prior success of heliox in the management of RDS combined with the recent advent of Hx-nCPAP we intend to investigate the utility of Hx-nCPAP in reducing the incidence of early nCPAP failure in ELBW infants with RDS.

Research design: Prospective, open-label, randomized, pilot study comparing conventional nCPAP to Hx-nCPAP in the management of ELBW infants being treated with nCPAP for RDS.

Methods: All spontaneously breathing infants born at < 30 wks estimated gestational age (EGA) admitted to the NICU at KMCWC with the diagnosis of RDS and on nCPAP since birth will be eligible for enrollment. Volunteer Infants will be randomly assigned to conventional nCPAP or Hx-nCPAP groups. Hx-nCPAP will be provided to the study group infants for the first 72 hours of life. Primary and secondary outcome measures will be compared between the heliox group and control group to determine if Hx-nCPAP results in a decreased incidence of early nCPAP failure and/or improved clinical outcomes when compared to conventional nCPAP.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 33 weeks
* Receiving CPAP from the time of delivery

Exclusion Criteria:

* Cyanotic congenital heart disease
* Congenital malformation

Ages: 1 Minute to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2008-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Nasal CPAP failure resulting in endotracheal intubation | 72 hours of life

SECONDARY OUTCOMES:
Bronchopulmonary dysplasia | 36 weeks corrected gestational age
Hospital length of stay | At hospital discharge
Death | Prior to hospital discharge
Pulmonary interstitial emphysema | 72 hours of life
Pneumothorax | 72 hours of life

CONTACTS AND LOCATIONS:
Overall Officials: Taylor Sawyer, DO, Study Director — Kapiolani Medical Center For Women & Children
Locations (1):
- Kapiolani Medical Center for Women and Children, Honolulu, Hawaii, United States